CLINICAL TRIAL: NCT01433796
Title: Tuberculosis in HIV-infected Patients Managed in Health Centres in Ethiopia - Identification of a Screening Algorithm for Active Tuberculosis and Determination of Outcome of Combined Antituberculosis and Antiretroviral Treatment
Brief Title: Screening for Tuberculosis in HIV-infected Patients Eligible for Antiretroviral Treatment
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Principal Investigator, Per Bjorkman, Associate professor, Lund University
Other Study IDs: LU-2010/672; 3120/215/03 (Other: Institute of Science and Technology, Ethiopia)
Record Dates: First submitted 2011-09-11; First posted 2011-09-14 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infection; Tuberculosis
Keywords: antiretroviral therapy; tuberculosis; health centres; Ethiopia
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aliquoted plasma samples from consenting participants are stored at -80 C for analysis of biomarkers of tuberculosis and for prognostic markers. Stool and urine samples are stored at -20 C for analysis of alternative biomarkers of active tuberculosis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Antiretroviral therapy, tuberculosis: Patients eligible for starting ART in health centres in Ethiopia

SUMMARY:
Background: Increased access to antiretroviral therapy (ART) in Africa will require decentralization to primary health care. For this purpose, adapted methods for management of patients co-infected with tuberculosis (TB) and HIV are needed. Improved detection of TB in patients starting ART, and assessment of co-administration of ART and TB treatment are priorities in this field.

Aims: To identify clinical predictors of TB in patients starting ART, and to construct screening algorithms for TB in this population; to assess ART outcomes in patients receiving TB treatment at health centre level.

Work plan: The project is performed in health centres providing ART in Ethiopia. A cohort of HIV positive patients initiating ART is prospectively followed. Baseline characteristics are registered; blood samples for CD4 cells, HIV RNA and immunological markers are collected, as well as sputum for TB culture and PCR. During ART, clinical data, CD4 cell counts and HIV RNA levels are followed. Patients with TB are compared to those without TB with regard to ART outcome. Baseline factors associated with TB will be used to construct TB screening algorithms.

Recruitment of the cohort was completed in March 2013; follow-up for determination of long term outcome of ART will be continued until 2016.

Significance: These studies give insight into TB-HIV co-infection at primary health care level in a Sub-Saharan region, and may impact future guidelines for management of such patients.

DETAILED DESCRIPTION:
Background: Tuberculosis (TB) remains as the leading opportunistic infection and cause of death among HIV-infected subjects in resource-limited settings (1). HIV infection is the strongest risk factor known for developing active TB, and as a consequence, the HIV epidemic in Sub-Saharan Africa has fuelled the incidence of TB (2). The interactions between HIV and TB are great challenges for health care, both with regard to diagnosis and treatment. In HIV-infected persons TB often has atypical manifestations, making correct and timely diagnosis difficult (3, 4). Recognition of TB before starting antiretroviral therapy (ART) is critical since a missed diagnosis of TB is associated with high early mortality after ART initiation (1, 5). Screening for TB is recommended for HIV-positive subjects, but a method with both satisfactory specificity and sensitivity that can be used in primary health care settings in Africa has not yet been identified. New diagnostic techniques for TB have recently been developed, such as the GenXpert PCR (6), but the optimal use of these alternative methods needs to be investigated.

In settings where both TB and HIV infection are common, a high proportion of patients are in need both of anti-tuberculosis treatment (ATT) and ART. Combined ART and ATT is associated with risks of drug interactions, overlapping side effects, immune reconstitution disease and poor adherence, but at least in patients with severe immunodeficiency, these risks are outweighed by decreased mortality (7-9). Studies performed in developed countries have shown that rates of virological suppression during ART in patients receiving concomitant ATT are comparable to those in persons not taking ATT (10, 11), but this topic has not been extensively investigated at primary health care level in Africa.

The number of HIV-infected subjects receiving ART in Sub-Saharan Africa has increased dramatically during the last years. Still, it is estimated that less than half of all patients in need of ART currently receive such treatment (12). In order to improve access, it will become necessary to further decentralize ART and to integrate this treatment into the primary health care system. Since many patients starting ART have unrecognized active TB at this time point, it is important to find a practical and reliable screening algorithm for TB among such individuals. Furthermore, the outcome of combined ATT and ART delivered in health centres must be assessed, especially with regard to HIV RNA suppression and selection of ART resistance.

This project aims to develop an algorithm with the potential to identify indicators of prevalent and incident TB among patients initiating ART by correlating baseline clinical signs and symptoms with results of culture- and PCR-based investigations for TB. Such clinical characteristics will be compared both to TB present before starting ART, as well as to TB presenting during the first year after ART initiation. Results from this comparison will be used to construct an algorithm for TB screening in Ethiopian patients eligible for ART. In addition, clinical, immunological and virological outcomes of ART in patients with concomitant ATT will be compared to those in patients only receiving ART. Specific aims are to study rates of virological suppression during ART, the development of antiretroviral drug resistance, and treatment adherence.

Work plan: HIV-infected adult patients eligible to start ART will be recruited from HIV clinics in several health centres providing integrated for HIV and TB in the Oromia region. 812 patients have been prospectively included into the cohort, and are under continued follow-up.

At baseline, detailed demographic, socio-economic and clinical data (such as presence of general and respiratory symptoms, body mass index, mid-upper arm circumference and various findings on physical examination) has been collected, including information on current medical and traditional therapies. Blood for CD4 cell count, complete blood count and HIV RNA will be obtained. In addition, plasma, stool and urine sample for analysis of immunological and inflammatory markers, and potential new biomarkers of active TB infection, has been collected and stored at -80 and -20 ° C.

Participants have undergone sampling for microbiological investigations for TB before starting ART. All patients have submitted two sputum samples for TB microscopy, culture and PCR. From patients with peripheral lymphadenopathy, lymph node aspiration for microbiological testing has been done. PCR has been performed using the GeneXpert technique. The study protocol will include definitions of TB based on microbiological results and clinical data according to WHO guidelines. Results of TB cultures are not awaited before ART initiation. Patients in whom TB is diagnosed receive ATT as soon as the diagnosis is established. For patients who have started ART at this time point, the recommendation will be to continue ART; however, the responsible clinician may decide to interrupt ART if medically indicated.

Follow up: Participants will be followed for 48 months (once monthly during the first 3 months, subsequently every 3 months for the first year of the study and then every 6 months). On follow-up visits, clinical and adherence data is collected. Incidence of death, hospitalization, TB and other opportunistic infections, signs of immune reconstitution inflammatory syndrome (IRIS), defaulting or treatment interruption is followed continuously, with tracing of defaulters to ascertain rates of mortality. Blood for CD4 cell counts and HIV RNA is obtained at 1 month after starting ART and at 3-monthly intervals for the first 6 months after study inclusion (and at 6-monthly intervals onwards). Samples obtained more than 6 months after starting ART with detectable HIV RNA will be subjected to genotypic testing to detect drug resistance mutations. In addition, blood samples for analysis of immunological markers will be obtained after 1, 3, 6 and 12 months of ART. Urine samples have been analyzed for the presence of lipoarabinomannane using a lateral flow assay.

Data analysis: Patient characteristics will be correlated with prevalent TB at baseline, to identify indicators of TB. These results will be used to construct screening algorithms that will be validated for sensitivity, specificity and predictive accuracy. Baseline predictors for incident TB during ART will also be investigated. For assessment of ART outcome, patients will be categorized according to their baseline TB status. Participants taking ATT will be compared to controls only taking ART. Incidence and time to defined events will be studied using survival curves (mortality, disease progression, HIV RNA suppression, loss to follow-up). HIV RNA and CD4 cell levels during ART, treatment interruptions, adherence, new opportunistic infections, drug side effects and TB IRIS will be compared between groups. Predictors of death and ART failure will be assessed.

Significance: Improving the management of patients co-infected with TB and HIV in highly endemic regions is critical for the success of continued scaling up of ART. Initiating ART during ATT is challenging under existing conditions in Sub-Saharan Africa, where the majority of these patients are diagnosed and treated. Case detection rates of TB remain below estimates in Ethiopia. Active TB is frequently missed in patients eligible for ART, a phenomenon likely to be important for mortality and medical complications following ART initiation. A screening algorithm based on clinical data with adequate predictive accuracy could help to identify TB in this population, and lead to improved treatment outcomes both for TB and HIV infection. Increased detection and timely treatment of TB in HIV-infected subjects would also reduce transmission in society. The outcome of combined ATT and ART administered in health centres must be assessed, especially concerning the development of drug resistance which can have serious consequences both for the infected individual and the community. Results from this study could inform health authorities on the efficacy and feasibility of such combined therapy, which is important for future HIV/TB policies in Ethiopia and other Sub-Saharan countries.

The project has received ethical clearance from Lund University, Sweden, and from the Institute of Science and Technology, Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Fulfills criteria for antiretroviral therapy (CD4 cell count below 350 cells/ml and/or WHO stage IV)
* Residence in study uptake area
* Written informed consent to participation and to tracing in case of defaulting

Exclusion Criteria:

* Ongoing or previous antiretroviral therapy
* Treatment for active tuberculosis for more than two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients managed in health centres
Sampling Method: Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Correlation between baseline clinical characteristics and presence of microbiologically confirmed active tuberculosis. | Two years
  To develop an algorithm with the potential to identify indicators of prevalent and incident TB among patients initiating ART by correlating baseline clinical signs and symptoms with results of culture- and PCR-based investigations for TB. Such clinical characteristics will be compared both to TB present before starting ART, as well as to TB presenting during the first year after ART initiation. Results from this comparison will be used to construct an algorithm for TB screening in Ethiopian patients eligible for ART.
Comparison of ART outcome in patients taking concomitant anti-tuberculosis therapy and those only taking ART. | Three years
  To prospectively compare clinical, immunological and virological outcomes of ART in patients with concomitant ATT to those in patients only receiving ART. Specific aims are to study rates of virological suppression during ART, the development of antiretroviral drug resistance, and treatment adherence.

SECONDARY OUTCOMES:
Comparison of diagnostic methods for detection of TB among HIV-infected subjects eligible to start ART. | Two years
  To compare the diagnostic yields of GeneXpert PCR, smear microscopy and novel tests for the detection of TB among HIV-infected subjects in Ethiopia eligible to start ART, using mycobacterial culture as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Per Björkman, M.D., Associate professor, Study Director — Lund University; Taye Tolera Balcha, M.D., Principal Investigator — Lund University; Erik Sturegård, M.D., Ph.D., Study Chair — Lund University; Patrik Medstrand, Professor, Study Chair — Lund University
Locations (5):
- Ethiopia (5):
  - Adama Health Centre, Ādama, Oromiya
  - Geda Health Centre, Ādama, Oromiya
  - Dhera Health Center, Dhera, Oromiya
  - Mojo Health Centre, Mojo, Oromiya
  - Welenchiti Health Centre, Welenchiti, Oromiya

REFERENCES:
- [Background] Lawn SD, Harries AD, Anglaret X, Myer L, Wood R. Early mortality among adults accessing antiretroviral treatment programmes in sub-Saharan Africa. AIDS. 2008 Oct 1;22(15):1897-908. doi: 10.1097/QAD.0b013e32830007cd. PMID 18784453
- [Background] World Health Organization. Global tuberculosis control: epidemiology, strategy, financing. WHO Report, 2009. Geneva: World Health Organization, 2009
- [Background] Wood R, Middelkoop K, Myer L, Grant AD, Whitelaw A, Lawn SD, Kaplan G, Huebner R, McIntyre J, Bekker LG. Undiagnosed tuberculosis in a community with high HIV prevalence: implications for tuberculosis control. Am J Respir Crit Care Med. 2007 Jan 1;175(1):87-93. doi: 10.1164/rccm.200606-759OC. Epub 2006 Sep 14. PMID 16973982
- [Background] Shah S, Demissie M, Lambert L, Ahmed J, Leulseged S, Kebede T, Melaku Z, Mengistu Y, Lemma E, Wells CD, Wuhib T, Nelson LJ. Intensified tuberculosis case finding among HIV-Infected persons from a voluntary counseling and testing center in Addis Ababa, Ethiopia. J Acquir Immune Defic Syndr. 2009 Apr 15;50(5):537-45. doi: 10.1097/QAI.0b013e318196761c. PMID 19223783
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Dean GL, Edwards SG, Ives NJ, Matthews G, Fox EF, Navaratne L, Fisher M, Taylor GP, Miller R, Taylor CB, de Ruiter A, Pozniak AL. Treatment of tuberculosis in HIV-infected persons in the era of highly active antiretroviral therapy. AIDS. 2002 Jan 4;16(1):75-83. doi: 10.1097/00002030-200201040-00010. PMID 11741165
- [Background] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray A, Gengiah T, Nair G, Bamber S, Singh A, Khan M, Pienaar J, El-Sadr W, Friedland G, Abdool Karim Q. Timing of initiation of antiretroviral drugs during tuberculosis therapy. N Engl J Med. 2010 Feb 25;362(8):697-706. doi: 10.1056/NEJMoa0905848. PMID 20181971
- [Background] Lawn SD, Myer L, Bekker LG, Wood R. Tuberculosis-associated immune reconstitution disease: incidence, risk factors and impact in an antiretroviral treatment service in South Africa. AIDS. 2007 Jan 30;21(3):335-41. doi: 10.1097/QAD.0b013e328011efac. PMID 17255740
- [Background] Breen RA, Miller RF, Gorsuch T, Smith CJ, Ainsworth J, Ballinger J, Swaden L, Cropley I, Johnson MA, Lipman MC. Virological response to highly active antiretroviral therapy is unaffected by antituberculosis therapy. J Infect Dis. 2006 May 15;193(10):1437-40. doi: 10.1086/503437. Epub 2006 Apr 4. PMID 16619192
- [Background] Hung CC, Chen MY, Hsiao CF, Hsieh SM, Sheng WH, Chang SC. Improved outcomes of HIV-1-infected adults with tuberculosis in the era of highly active antiretroviral therapy. AIDS. 2003 Dec 5;17(18):2615-22. doi: 10.1097/00002030-200312050-00008. PMID 14685055
- [Background] Towards universal access: scaling up priority HIV/AIDS interventions in the health sector. September 2009 progress report. WHO 2009
- [Derived] Balcha TT, Skogmar S, Sturegard E, Schon T, Winqvist N, Reepalu A, Jemal ZH, Tibesso G, Bjork J, Bjorkman P. A Clinical Scoring Algorithm for Determination of the Risk of Tuberculosis in HIV-Infected Adults: A Cohort Study Performed at Ethiopian Health Centers. Open Forum Infect Dis. 2014 Oct 10;1(3):ofu095. doi: 10.1093/ofid/ofu095. eCollection 2014 Dec. PMID 25734163
- [Derived] Reepalu A, Balcha TT, Skogmar S, Jemal ZH, Sturegard E, Medstrand P, Bjorkman P. High rates of virological suppression in a cohort of human immunodeficiency virus-positive adults receiving antiretroviral therapy in ethiopian health centers irrespective of concomitant tuberculosis. Open Forum Infect Dis. 2014 Jun 19;1(1):ofu039. doi: 10.1093/ofid/ofu039. eCollection 2014 Mar. PMID 25734107
- [Derived] Reepalu A, Balcha TT, Skogmar S, Jemal ZH, Sturegard E, Medstrand P, Bjorkman P. High rates of viral suppression in a cohort of HIV-positive adults receiving ART in Ethiopian health centers irrespective of concomitant tuberculosis. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19612. doi: 10.7448/IAS.17.4.19612. eCollection 2014. PMID 25394116
- [Derived] Balcha TT, Sturegard E, Winqvist N, Skogmar S, Reepalu A, Jemal ZH, Tibesso G, Schon T, Bjorkman P. Intensified tuberculosis case-finding in HIV-positive adults managed at Ethiopian health centers: diagnostic yield of Xpert MTB/RIF compared with smear microscopy and liquid culture. PLoS One. 2014 Jan 22;9(1):e85478. doi: 10.1371/journal.pone.0085478. eCollection 2014. PMID 24465572